CLINICAL TRIAL: NCT06216912
Title: Ultrasound Assessment of Gastric Volume in Paralyzed Obese Patients After High-flow Nasal Oxygen Therapy
Brief Title: Gastric Volume in Paralyzed Obese Patients After High-flow Nasal Oxygen Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HFNOT_gastric
Record Dates: First submitted 2024-01-03; First posted 2024-01-22 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-01

CONDITIONS: Undefined

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative preoxygenation is performed using High-flow nasal oxygen therapy, and the gastric volume before and after High-flow nasal oxygen therapy is measured by ultrasound and compared in obese patients undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
Preoperative preoxygenation is performed using High-flow nasal oxygen therapy, and the gastric volume before and after High-flow nasal oxygen therapy is measured by ultrasound and compared in obese patients undergoing surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a BMI of 30 kg/m2 or more, undergoing surgery under general anesthesia

Exclusion Criteria:

* Nasotracheal intubation
* History of a surgery or anatomical anomaly in the head and neck
* History of Inability to breathe through nose
* History of difficult airway
* Severe cardiac or respiratory disease
* Gastric reflux disease, diabetes, pregnancy
* Previous gastric surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients undergoing surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
gastric volume measured by gastric ultrasound | immediately before HFNOT, immediately after HFNOT, immediately after tracheal intubation
  gastric volume measured by gastric ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- SMG - SNU Boramae Medical Center, Seoul, South Korea